CLINICAL TRIAL: NCT05642325
Title: A Phase III, Multicenter, Randomized, Double-Masked, Sham-Controlled Study to Investigate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Vamikibart Administered Intravitreally in Patients With Uveitic Macular Edema
Brief Title: Vamikibart in Participants With Uveitic Macular Edema
Acronym: Sandcat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GR44278; 2022-501794-39-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-06; First posted 2022-12-08 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Uveitic Macular Edema
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Participants will receive 4 high-dose vamikibart intravitreal (IVT) injections every 4 weeks (Q4W) to Week 12, followed by as-needed (PRN) dosing from Week 20 to Week 48.
  Interventions: Drug: Vamikibart
- Arm B (Experimental): Participants will receive 4 low-dose vamikibart IVT injections Q4W to Week 12, followed by PRN dosing from Week 20 to Week 48.
  Interventions: Drug: Vamikibart
- Arm C (Sham Comparator): Participants will receive 4 sham injections Q4W to Week 12, followed by PRN sham dosing from Week 20 to Week 48.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Vamikibart — Participants will receive vamikibart IVT injection
  Other Names: RO7200220
  Arms: Arm A; Arm B
Other: Sham — Participants will receive a sham procedure that mimics an IVT injection.
  Arms: Arm C

SUMMARY:
This study will assess the efficacy and safety of vamikibart in participants with uveitic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Female participants: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception as defined by the protocol
* Diagnosis of macular edema associated with non-infectious uveitis (NIU)
* Diagnosis of active or inactive, acute, or chronic NIU of any etiology and of any anatomical type (anterior, intermediate, posterior, panuveitis)
* BCVA letter score of 73 to 19 letters (inclusive) on Early Treatment Diabetic Retinopathy Study (EDTRS)-like charts

Exclusion Criteria:

* Evidence of active or latent syphilis infection
* Evidence of active or latent tuberculosis infection and/or positive tuberculosis assay, or previous or current HIV diagnosis
* Serious acute or chronic medical or psychiatric illness
* History of major ocular and non-ocular surgical procedures
* Uncontrolled IOP or glaucoma or chronic hypotony
* Any anatomical changes or media opacity in the study eye preventing evaluation of retina, vitreous, and capture of study images
* Prior use of IVT biologics including anti-VEGFs less than 2-4 months prior to Day 1; received IVT Methotrexate within 4 months prior to Day 1
* Prior macular laser therapy, cataract surgery within 6 months and laser capsulotomy within 3 months of Day 1
* Topical corticosteroids and/or topical NSAID > 3 drops per day in the 14 days prior to Day 1 (D1); intraocular or periocular corticosteroid injections in the 2 months prior to D1; subconjunctival corticosteroid injection within 1 month prior to Day 1; an OZURDEX implant in the 4 months prior to D1; YUTIQ, RETISERT or ILUVIEN implant in the 3 years prior to D1
* Diagnosis of macular edema due to any cause other than NIU
* Any major ocular conditions that may require medical or surgical intervention during the study period to prevent vision loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with ≥ 15 letter improvement from baseline in best-corrected visual acuity (BCVA) at Week 16 | Week 16

SECONDARY OUTCOMES:
Proportion of participants with ≥ 15 letter improvement from baseline in BCVA at Week 20 | Week 20
Change from baseline in BCVA at Week 16 | Week 16
Change from baseline in central subfield thickness (CST) at Week 16 | Week 16
Change from Baseline in BCVA at Weeks 20 and 52 | Weeks 20 and 52
Change from baseline in CST at Weeks 20 and 52 | Weeks 20 and 52
Proportion of participants with uveitic macular edema secondary to non-infectious uveitis (UME) resolution defined by standardized (by machine) CST threshold <325um on optical coherence tomography (OCT) from baseline at Weeks 16 and 52 | Weeks 16 and 52
Time to rescue treatment | Up to Week 52
Number of rescue treatments received | Up to Week 52
Type of rescue treatments received | Up to Week 52
Proportion of participants with ≥15 letter improvement from baseline in BCVA at Week 16 and 52 | Weeks 16 and 52
Proportion of participants without ≥15 letter loss from baseline in BCVA at Week 16 and 52 | Weeks 16 and 52
Time to first PRN injection | Up to Week 52
Change from baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) at Weeks 16 and 52 | Weeks 16 and 52
Percentage of participants with ocular adverse events (AEs) | Up to Week 52
Percent change from baseline in corneal endothelial cell density at Week 24 | Week 24
Percentage of participants with non-ocular AEs | Up to Week 52
Percentage of participants with adverse events of special interest (AESIs) | Up to Week 52
Percent change from baseline in corneal endothelial cell density at Week 52 | Week 52
Aqueous humor (AH) concentration of vamikibart | Up to Week 52
Serum concentration of vamikibart | Up to Week 52
Anti-drug antibody titer to vamikibart | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (94):
- United States (23):
  - Associated Retina Consultants, Phoenix, Arizona
  - Barnet Dulaney Perkins Eye Center, Sun City, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - California Eye Specialists Medical group Inc., Pasadena, California
  - Retina Consultants of Southern California, Redlands, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - University of California, Davis, Eye Center, Sacramento, California
  - Retinal Consultants Med Group, Sacramento, California
  - Advanced Research, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Duke Eye Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Erie Retina Research, Erie, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Retina Group of Washington, Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Argentina (5):
  - Centro Privado de Ojos, Ciudad Autonoma Buenos Aires
  - Buenos Aires Mácula, Ciudad Autonoma Buenos Aires
  - Consultorios Medicos Oftalmológicos, Ciudad Autonoma Buenos Aires
  - Oftalmologia Global, Rosario
  - Organizacion Medica de Investigacion, San Nicolás
- Australia (5):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Eye Surgery Associates, Malvern, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
- General Teaching Hospital Prague, Prague, Czechia
- France (4):
  - CHU Nantes - Hotel Dieu, Nantes
  - Hopital Lariboisiere, Paris
  - Hôpital COCHIN, Paris
  - Ch Pitie Salpetriere, Paris
- Germany (10):
  - Charité-Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin
  - Universitatsklinikum Koln, Cologne
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinik Heidelberg, Heidelberg
  - Universitätskliniikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - St. Franziskus Hospital, Münster
  - Knappschaftsklinikum Saar GmbH, Sulzbach
  - Universitäts-Augenklinik Tübingen, Tübingen
- India (5):
  - Narayana Nethralaya Hospital, Bangalore, Karnataka
  - Sankara Nethralaya, Chennai, Tamil Nadu
  - L V Prasad Eye Institute, Hyderabad, Telangana
  - ICARE Eye Hospital & PG Institute, Noida, Uttar Pradesh
  - Postgraduate Institute of Medical Education and Research, Chandigarh
- Italy (3):
  - AUSL ? IRCCS Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Asst Fatebenefratelli Sacco, Milan, Lombardy
- Japan (14):
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Hokkaido University Hospital, Hokkaido
  - Kobe University Hospital, Hyōgo
  - Kagoshima University Hospital, Kagoshima
  - Yokohama City University Hospital, Kanagawa
  - Japan Community Health care Organization Osaka Hospital, Osaka
  - The University of Osaka Hospital, Osaka
  - Jichi Medical University Saitama Medical Center, Saitama
  - National Defense Medical College Hospital, Saitama
  - Tokyo Medical University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
  - Nippon Medical School Tama Nagayama Hospital, Tokyo
  - Yamaguchi University Hospital, Yamaguchi
- "Kazakh "Badge of H?nour" Scientific R?s??r?h Institute of ??? diseases" LLP, Almaty, Kazakhstan
- Portugal (2):
  - AIBILI - Association for Innovation and Biomedical Research on Light, Coimbra
  - Hospital de Santa Maria, Lisbon
- National University Hospital, Singapore, Singapore
- South Korea (3):
  - Pusan National University Hospital, Busan
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (5):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Clinic Barcelona, Barcelona
  - Fundacion Jimenez Diaz-UTE, Madrid
  - Hospital Clinico San Carlos, Madrid
- Switzerland (4):
  - Inselspital Bern Ophthalmologische Klinik, Bern
  - Berner Augenklinik, Bern
  - Vista Klinik Ophthalmologische Klinik, Binningen
  - Stadtspital Triemli Ophthalmologische Klinik, Zurich
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Ege Üniversitesi Tip Fakültesi, Lzmir
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing